CLINICAL TRIAL: NCT03386942
Title: A Phase 1 Study of MORAb-202 in Subjects With Solid Tumors
Brief Title: A Study of MORAb-202 (Herein Referred to as Farletuzumab Ecteribulin) in Participants With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MORAb-202-J081-101
Record Dates: First submitted 2017-11-28; First posted 2017-12-29 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Solid Tumors
Keywords: Solid Tumors; Folate Receptor α (FRA) and platinum-resistant ovarian carcinoma; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Pyogenic arthritis, pyoderma gangrenosum, and acne; Carcinoma, Non-Small-Cell Lung | interventions — MORAb-202

STUDY DESIGN:
Intervention Model Description: This is a Phase 1 study of farletuzumab ecteribulin in participants with solid tumors. This study will be conducted in 2 parts (Part 1 and Part 2). Part 1 will be the dose escalation portion of this study to evaluate dose-limiting toxicity (DLT) and to determine the maximum tolerated dose (MTD) of farletuzumab ecteribulin in participants with solid tumors. Considering efficacy, safety, and the pharmacokinetic (PK) profile, two doses may be selected from Part 1 for Part 2. Part 2 will comprise cohort expansions to further characterize the safety of farletuzumab ecteribulin and to evaluate the preliminary efficacy of farletuzumab ecteribulin in participants with FRA-positive platinum-resistant ovarian carcinoma and non-small cell lung cancer (NSCLC). The recommended dose for future studies will be determined based on the data from Part 1 and Part 2.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Farletuzumab Ecteribulin (Experimental): Part 1 (Dose-escalation): The initial dose level of farletuzumab ecteribulin will be 0.3 milligrams per kilogram (mg/kg) every 3 weeks in the first cohort with 1 participant for dose-limiting toxicity (DLT) evaluation. DLTs will be evaluated in successive dose level cohorts with a single participant until a drug-related Grade 2 or higher toxicity is observed. If such a toxicity is observed, the cohort will be expanded to enroll a total of 3 participants.
  Part 2 (Treatment Phase): farletuzumab ecteribulin will be administered every 3 weeks during the treatment phase at the dose determined in Part 1 until participants meet any of the criteria for discontinuation. Criteria for discontinuation include: withdrawal of consent, major protocol violations, unable to continue due to adverse events, pregnancy, progressive disease, Investigator decision, or infusion reactions.
  Interventions: Drug: Farletuzumab Ecteribulin

INTERVENTIONS:
Drug: Farletuzumab Ecteribulin — Part 1: farletuzumab ecteribulin intravenous (IV) infusion administered every 3 weeks starting at a 0.3 mg/kg dose and successively increasing doses until DLT. Part 2: farletuzumab ecteribulin administered IV every 3 weeks at a dose determined in Part 1 until any of the criteria for discontinuation are met.
  Other Names: MORAb-202

SUMMARY:
The primary objective of this study is to evaluate the tolerability and safety profile of farletuzumab ecteribulin in participants with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have provided voluntary written consent for participation in this clinical study.
* Participants to whom the rules for complying with this clinical study have been adequately explained, and who intend to and can comply with those rules.
* Male or female participants age >=20 years at the time of informed consent of screening 1 (or screening 2, in case of participants who enter this clinical study from screening 2).
* Part 1 only: Participants with FRA-positive solid tumor confirmed by immunohistochemistry (IHC) assay at the central laboratory using their available tumor samples from resected specimen (i.e., surgical or excisional/incisional biopsy samples) or core needle biopsy (<=18-gauge), or participants with a histological and/or cytological diagnosis of any serous ovarian carcinoma, fallopian tube carcinoma, endometrial carcinoma, or adenocarcinoma of Non-Small Cell Lung Cancer (NSCLC), whose archival resected tumor samples (that is, surgical or excisional/incisional biopsy sample).
* Part 1 only: At informed consent of screening 2, participants who failed standard therapies, or for which no appropriate treatment is available.
* Participants with adequate function of major organs within 2 weeks prior to the first administration of the study drug as follows.

  1. Hemoglobin >=9.0 grams per deciliter (g/dL).
  2. Neutrophil count >=1.5 × 10^3/microliters (μL).
  3. Platelet count >=10 × 10^4/μL.
  4. Total bilirubin <=1.5 × upper limit of normal (ULN) in the facility.
  5. Alanine aminotransferase and aspartate aminotransferase <=3.0 × ULN in the facility (in the case of liver metastases <=5*ULN).
  6. Serum creatinine <=1.5 × ULN in the facility.
  7. Albumin >=3 g/dL.
* Participants with Performance Status score of 0-1 established by Eastern Cooperative Oncology Group.
* Participants who are expected to survive for 3 months or longer after the first administration of the study drug.
* Washout period required from the end of prior treatment to the first administration of the study drug will be as follows

  a. Anticancer therapy
  * Antibody and other study drugs: >4 weeks (however, in the case where the half-life of other study drugs is known and 5 × half-lives of that study drug is less than or equal to 4 weeks, participants can be eligible after >=5 × half-lives of that study drug has passed).
  * Prior chemotherapy (except small-molecule targeted therapy), surgical therapy, radiation therapy: >3 weeks.
  * Endocrine therapy, immunotherapy except antibody, small-molecule targeted therapy: >2 weeks.
* Supportive therapies

  • Blood/platelet transfusion, hematopoietic stimulating agent including granulocyte colony-stimulating factor formulation: > 2 weeks.
* Participants whose formalin fixed, paraffin-embedded unstained slides of tumor sample are available for IHC test at central laboratory. If applicable biopsy will be performed by excisional, incisional or needle puncture (<=18-gauge as far as possible).

Inclusion Criteria (Part 2 only)

* Measurable disease meeting the following criteria:

  1. At least 1 lesion of >=1.0 centimeters (cm) in the longest diameter for a non-lymph node or >=1.5 cm in the short-axis diameter for a lymph node that is measurable according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 using computerized tomography/magnetic resonance imaging.
  2. Lesions that have had external beam radiotherapy or locoregional therapies such as radiofrequency ablation must show evidence of progressive disease based on RECIST 1.1 to be deemed a target lesion.
* Participants histologically diagnosed with the following ovarian carcinoma (including primary peritoneal carcinoma and fallopian tube carcinoma) or NSCLC. Participants for Cohort 1 and 3 who have archival resected tumor samples (that is, surgical or excisional/incisional biopsy sample) for IHC assay are not required to be FRA positive at the central laboratory (Screening 1 is not required). Participants for Cohort 1 and 3 who do not have archival resected tumor samples (that is, surgical or excisional/incisional biopsy sample) are required to be FRA positive at the central laboratory (Screening 1 is required). Participants for Cohort 2 and 4 are required to be FRA positive confirmed by IHC assay at the central laboratory using their available tumor samples from resected specimen (that is, surgical or excisional/incisional biopsy samples) or core needle biopsy (<=18-gauge for ovarian carcinoma and for NSCLC [adenocarcinoma and non-adenocarcinoma] as possible) (Screening 1 is required).

  * Cohort 1: High grade serous adenocarcinoma
  * Cohort 2: Other histological types of ovarian carcinoma (excluding mucinous adenocarcinoma)
  * Cohort 3: NSCLC adenocarcinoma
  * Cohort 4: NSCLC non-adenocarcinoma
* Participants with the following disease characteristics:

  1. Ovarian carcinoma (including primary peritoneal carcinoma and fallopian tube carcinoma):

     * Participants with platinum-resistant disease (defined as progression radiographically within less than [<] 6 months from completion of last platinum therapy) who have received >4 cycles in last platinum-containing chemotherapy for ovarian carcinoma
     * Participants who have received up to two regimen of chemotherapy after diagnosed as platinum-resistant
  2. NSCLC:

     * Participants that have advanced after previous treatment and those for which no alternative standard therapy exist and those who are not indicated for epidermal growth factor receptor (EGFR), BRAF V600E mutation, anaplastic lymphoma kinase (ALK) or reactive oxygen species (ROS)-targeted therapy (Participants who have progressed after prior such therapy may be eligible)

Exclusion Criteria:

* Medical history of clinically significant cardiovascular impairment:

  1. Congestive heart failure greater than or equal to New York Heart Association Class III.
  2. Unstable angina pectoris, myocardial infarction or stroke within 6 months before of the first administration of the study drug.
  3. Prolongation of corrected QT (QTc) interval to > 480 milliseconds (ms) (Fridericia method).
  4. Arrhythmias associated with hemodynamic instability.
* Concomitant systemic infection requiring medical treatment.
* Participants who test positive for human immunodeficiency virus (HIV antibody).
* Active viral hepatitis (B or C) (*) as demonstrated by positive serology or requiring treatment.

(*) hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (anti-HBs)/hepatitis B core antibody (HBcAb), and anti-hepatitis C virus (HCV) antibody test. Participants who are anti-HBs/HBcAb (+) without detectable hepatitis B virus (HBV)-deoxyribonucleic acid (DNA)/HCV- ribonucleic acid (RNA) are eligible.

* Effusion requiring drainage continually.
* Participants whose toxicity of previous treatment has not recovered to Grade 1 or lower (except for alopecia and hemoglobin).
* Participants who have received a previous monoclonal antibody therapy and have evidence of an immune or allergic serious reaction.
* Participants who had previous treatment with other folate receptor targeting agents.
* Participants who have medical history of discontinuing prior eribulin due to toxicity.
* Has an active pneumonitis/interstitial lung disease (ILD), a history of pneumonitis/ILD that required systemic steroids, received radiotherapy to lung field within 12 months before the first dose of study intervention, or current clinically relevant lung disease (example, Chronic Obstructive Pulmonary Disease).
* Other active malignancy (except for definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix) within the past 24 months prior to the first administration of the study drug.
* Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin or human chorionic gonadotropin). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 3 days before the first administration of the study drug (breastfeeding participants are not eligible even if they discontinue breastfeeding).
* Women of childbearing potential or man of impregnate potential who don't agree that both the participant and his/her partner will use a medically effective method for contraception (as below) during the study and after study drug discontinuation (male; 90 days, female; 60 days).

Note: Condom*, contraceptive sponge**, foam**, jelly**, diaphragm*, intrauterine device*, or use of oral contraception* from at least 4 weeks before starting the study treatment (*Approved drugs or certified medical devices in Japan, **Non-approved drugs or certified medical devices in Japan).

* Known intolerance to the study drug or any of the excipients.
* Any medical or other condition that in the opinion of the investigator(s) would preclude the participant's participation in the study.
* Scheduled for surgery during the study.
* Diagnosed with meningeal carcinomatosis.
* Participants with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment in this study. Any signs (e.g., radiologic) or symptoms of brain metastases must be stable for at least 4 weeks before starting study treatment.
* Use of illegal recreational drugs.

Exclusion Criteria (Part 2 only)

* Previous treatment with eribulin
* Participants histologically diagnosed with mucinous ovarian carcinoma
* (Ovarian carcinoma only) Participants who progressed during the preceding platinum-containing chemotherapy (for platinum refractory)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of participants with dose-limiting toxicities (DLTs) | At the end of Cycle 1 (21 days)
  DLTs are defined as the following occurring in Cycle 1 for which a causal relationship with study drug cannot be ruled out: febrile neutropenia, Grade 4 neutropenia persisting for more than 7 days, or neutropenia requiring hematopoietic stimulating agents, Grade 4 thrombocytopenia, or thrombocytopenia requiring platelet transfusion, Grade 4 anemia, or anemia requiring blood transfusion, Grade 3 non-hematological toxicity (except abnormal clinical laboratory values of no clinical significance, any events which can be managed and controlled to Grade 2 or less by maximal medical management, infusion reactions of Grade 3 or higher are NOT considered DLTs because they are stochastic and idiosyncratic events, not related to dose), Grade 4 non-hematological toxicity, and/or when the second treatment with farletuzumab ecteribulin is postponed more than 14 days from the scheduled day due to toxicity. DLTs will be determined by discussion between the investigator, sponsor, and medical expert.
Part 1 and Part 2: Number of participants with adverse events (AEs), adverse events of interest (AEIs), and serious adverse events (SAEs) | Up to 50 months
Number of participants with any clinically significant clinical laboratory test value | Up to 50 months
  Clinical significance will be determined by the Investigator.
Number of participants with any clinically significant vital sign value | Up to 50 months
  Clinical significance will be determined by the Investigator.
Change from Baseline in arterial oxygen saturation | Baseline; up to 50 months
Change from Baseline in body weight | Baseline; up to 50 months
Number of participants with any clinically significant 12-lead electrocardiogram (ECG) value | Up to 50 months
  Clinical significance will be determined by the Investigator.
Change from Baseline in the performance status (PS) score established by the Eastern Cooperative Oncology Group (ECOG) | Baseline; up to 50 months
Change from Baseline in serum anti-drug antibody (ADA) titer | Baseline; up to 50 months

SECONDARY OUTCOMES:
Part 1: Maximum Tolerated Dose (MTD) of Farletuzumab Ecteribulin | 21 days following each dose level of farletuzumab ecteribulin (up to a maximum of 50 months)
  The MTD will be selected as the dose with the smallest difference between the target DLT rate of 25% and an estimate of DLT rate based on the posterior distribution of DLT rate for each dose.
Part 1 and Part 2: Maximum observed serum concentration (Cmax) of Farletuzumab Ecteribulin | Predose; end of infusion; 0.5, 1, 2, 4, and 24 hours post infusion on Day 1; on Days 4, 8, and 15; and the discontinuation and last observation visit (up to 50 months)
  Cmax is the maximum serum concentration of farletuzumab ecteribulin after administration of the drug.
Part 1 and Part 2: Maximum serum concentration of total antibody | Predose; end of infusion; 0.5, 1, 2, 4, and 24 hours post infusion on Day 1; on Days 4, 8, and 15; and the discontinuation and last observation visit (up to 50 months)
Part 1 and Part 2: Plasma concentration of free eribulin | Predose; end of infusion; 0.5, 1, 2, 4, and 24 hours post infusion on Day 1; on Days 4, 8, and 15; and the discontinuation and last observation visit (up to 50 months)
Recommended dose (RD) of farletuzumab ecteribulin for future studies | From the date of screening until the last observation visit (up to 50 months)
  The RD will be determined based on the MTD, efficacy, and safety data in Part 1 and Part 2.
Part 1 and Part 2: Best overall response (BOR) | From the date of screening until the last observation visit (up to 50 months)
  BOR was based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). BORs are complete response (CR), partial response (PR), stable disease (SD), progression of disease (PD), and not evaluable (NE), where SD has to be achieved at ≥5 weeks after the first dose. CR or PR in Part 1 of this study requires no confirmation of the next response at ≥4 weeks. CR or PR in Part 2 of this study requires confirmation of the next response at ≥4 weeks.
Part 1 and Part 2: Overall response rate (ORR) | From the date of screening until the last observation visit (up to 50 months)
  ORR is defined as the percentage of participants with BOR of CR or PR.
Part 1 and Part 2: Disease control rate (DCR) | From the date of screening until the last observation visit (up to 50 months)
  DCR is defined as the percentage of participants with BOR of CR, PR, or SD.
Part 1 and Part 2: Clinical benefit rate (CBR) | From the date of screening until the last observation visit (up to 50 months)
  CBR is defined as the percentage of participants with BOR of CR, PR or durable (SD) (duration of SD ≥ 23 weeks).
Part 2: Duration of Response (DOR) | From the date of screening until the last observation visit (up to 50 months)
  DOR is defined as the time from the first documentation of CR or PR to the first documented date of event (disease progression or death from any cause, whichever occurs first).
Part 2: Progression-free survival (PFS) | From the date of screening until disease progression or death (up to 50 months)
  PFS is defined as the time from the date of the first dose of study drug to the first documented date of event (disease progression or death from any cause, whichever occurs first).
Part 2: Overall Survival (OS) | From the date of screening until the last observation visit (up to 50 months)
  OS is defined as the time from the date of the first dose to the date of death from any cause. For participants who are alive or unknown, OS is censored as the date of the last known alive date or the date of data cut off, whichever comes first.

CONTACTS AND LOCATIONS:
Locations (10):
- Japan (10):
  - Eisai Trial Site 5, Matsuyama, Ehime
  - Eisai Trial Site 6, Kurume, Fukuoka
  - Eisai Trial Site 8, Sapporo, Hokkaido
  - Eisai Trial Site 4, Akashi, Hyōgo
  - Eisai Trial Site 7, Niigata, Niigata
  - Eisai Trial Site 3, Hidaka, Saitama
  - Eisai Trial Site 9, Sunto-gun, Shizuoka
  - Eisai Trial Site 1, Chuo-ku, Tokyo
  - Eisai Trial Site 10, Koto-Ku, Tokyo
  - Eisai Trial Site 2, Koto-ku, Tokyo

REFERENCES:
- [Derived] Yonemori K, Yunokawa M, Matsumoto K, Takehara K, Hasegawa K, Hirashima Y, Kato H, Ikezawa H, Otake Y, Yusa W, Miura T, Nishio S. Clinical trial of safety and antitumor activity of farletuzumab ecteribulin in patients with platinum-resistant ovarian cancer: Phase I expansion results. Int J Gynaecol Obstet. 2025 Dec 23. doi: 10.1002/ijgo.70676. Online ahead of print. PMID 41432226
- [Derived] Shimizu T, Fujiwara Y, Yonemori K, Koyama T, Sato J, Tamura K, Shimomura A, Ikezawa H, Nomoto M, Furuuchi K, Nakajima R, Miura T, Yamamoto N. First-in-Human Phase 1 Study of MORAb-202, an Antibody-Drug Conjugate Comprising Farletuzumab Linked to Eribulin Mesylate, in Patients with Folate Receptor-alpha-Positive Advanced Solid Tumors. Clin Cancer Res. 2021 Jul 15;27(14):3905-3915. doi: 10.1158/1078-0432.CCR-20-4740. Epub 2021 Apr 29. PMID 33926914